CLINICAL TRIAL: NCT06339385
Title: Management of Pain, Agitation-sedation, Delirium Immobility and Sleep Disruption in Emergency Intensive Care Unit: a Multicenter Cross-sectional Survey
Brief Title: Management of PADIS in Emergency Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Collaborators: Beijing Tiantan Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Fudan University (Other); Affiliated hospital of Guilin medical university,China (Unknown); The Second Affiliated Hospital of Hainan Medical University (Other); The First Hospital of Hebei Medical University (Other); The First Hospital of Jilin University (Other); Southwest Hospital, China (Other); General hospital of shenyang military command (Unknown); Beijing Anzhen Hospital (Other); Mianyang Central Hospital (Other); Tianjin Medical University General Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); The Jiangxi Provincial People's Hospital (Unknown)
Responsible Party: Principal Investigator, Zhou Yi-Min, Principal Investigator, Capital Medical University
Other Study IDs: KY 2020-153-02
Record Dates: First submitted 2024-03-25; First posted 2024-04-01 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Pain; Agitation, Emergence; Delirium; Critical Illness
Keywords: Emergency Department Intensive Care Units; Prevalence; Survey; Practices
MeSH Terms: conditions — Pain; Emergence Delirium; Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EDICU patients: All patients admitted to the participating EDICU during the on-site investigation.
  Interventions: Behavioral: PADIS assessment

INTERVENTIONS:
Behavioral: PADIS assessment — Hospital and nursing records from the 24 hours preceding enrollment were examined to document the assessment rate of pain, agitation-sedation, and delirium.

SUMMARY:
Investigate the prevalence of PADIS in EICU, as well as the awareness and clinical implementation status of medical staff towards PADIS.

The investigators conducted a multicenter cross-sectional survey in mainland China, including a one-day point prevalence investigation and a questionnaire survey. The inclusion criteria encompassed all adult patients admitted to the participating emergency department intensive care units (EDICUs) during the on-site screening, while exclusion criteria comprised patients aged less than 18 years, EDICU stays duration less than 24 hours before the screening, and participation in other concurrent trials. Hospital and nursing records from the 24 hours preceding enrollment were examined to document the assessment rate of pain, agitation-sedation, and delirium. Physicians and nurses on duty 24 hours before the patients' enrollment was invited to complete the questionnaire survey regarding the ICU profiles, professional expertise, assessment and treatment of PAD, early mobilization, and sleep improvement practices.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the participating EDICU during the on-site investigation

Exclusion Criteria:

* Age less than 18 years;
* EDICU stay duration before the screening was less than 24 hours
* Enrollment in other concurrent trials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to the participating EDICU during the on-site investigation were eligible for enrollment in this study. However, patients meeting the following criteria were excluded: 1) age less than 18 years; 2) EDICU stay duration before the screening was less than 24 hours; 3) enrollment in other concurrent trials.
Sampling Method: Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2021-06-13 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
PADIS assessment rate | 24 hours before enrollment

SECONDARY OUTCOMES:
Rates of analgesic and sedative administration | 24 hours before enrollment
Rate of accidental removal of the catheter during the EICU stay | From the start of the survey day until transfer out of the EDICU or 60 days after the survey day.
EDICU length of stay | From the start of the survey day until transfer out of the EDICU or 60 days after the survey day.
The hospital length of stay | From the start of the survey day until transfer out of the EDICU or 60 days after the survey day.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No